CLINICAL TRIAL: NCT04304066
Title: Research for the Molecular Imaging of the PD-L1 Targeting Tracer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019KT116/2019KT62
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging cohort (Experimental): All study participants will be allocated to this arm (single-arm study).Study participants will undergo 18F-WL12 or 68Ga-WL12 PET/CT scans
  Interventions: Other: 18F-WL12 PET or 68Ga-WL12 PET

INTERVENTIONS:
Other: 18F-WL12 PET or 68Ga-WL12 PET — WL12, labeled with PET radio-nuclide ( Ga-68 or F-18)will be used as a molecular imaging tracer for PET/CT scanning

SUMMARY:
To use the molecular probe PET radionuclide (Ga-68 or F-18) WL12 peptide to detect the expression of PD-L1 in the primary and metastatic lesions in patients with solid tumor; to detect the expression heterogeneity of PD-L1 in the lesion and inter-lesions; to observe the change of PD-L1 expression in the course of treatment. To provide an approach for screening patients with high expression of PD-L1, efficacy monitoring, drug resistance and early warning of recurrence and metastasis to achieve the Individualized antitumor treatment of targeted drugs.

DETAILED DESCRIPTION:
In many clinical trials, Anti-PD-1/PD-L1 mAbs have achieved great success than expected in a variety of refractory and recurrent tumor patients. The latest research shows that it is not all cancer patients would respond to Anti-PD-1/PD-L1 mAbs. At present, immunohistochemistry (IHC) is still a common method to screen patients that will benefit from this therapy by detecting the expression level of PD-1 and PD-L1. However, the results of IHC were not very exact because of limitations of IHC such as the heterogeneity of expression, the influence of host cell PD-L1 expression and the changes in the course of the disease. Moreover, the tumor tissue used in IHC must obtained through the invasive method. It is difficult to dynamically monitor the expression level of PD-1 / PD-L1 during the treatment. Immuno-PET molecular imaging By radiolabeling Anti-PD-1/PD-L1 mAbs with radionuclides can be used to noninvasive assessment of biodistribution of monoclonal antibodies and provide a new strategy for patient screening.

In this study, 18F-WL12 or 68Ga-WL12 PET / CT imaging will be performed in patients with solid tumors to access the potential of 18F-WL12 or 68Ga-WL12PET / CT to screen patients who can benefit from JS001 treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged >18 years old; ECoG 0 or 1;
* 2. Patients with solid tumors;
* 3. Has at least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST V1.1);
* 4. life expectancy >=12 weeks.

Exclusion Criteria:

* 1. Significant hepatic or renal dysfunction;
* 2. Is pregnant or ready to pregnant;
* 3. Cannot keep their states for half an hour;
* 4. Refusal to join the clinical study;
* 5. Suffering from claustrophobia or other mental diseases;
* 6. Any other situation that researchers think it is not suitable to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
SUV | 2 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value（SUV）on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Shunlian Zhou, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou X, Yan S, Li D, Zhu H, Liu B, Liu S, Zhao W, Yang Z, Wu N, Li N. Radiolabelled anti-PD-L1 peptide PET/CT in predicting the efficacy of neoadjuvant immunotherapy combined with chemotherapy in resectable non-small cell lung cancer. Ann Nucl Med. 2025 Apr;39(4):364-372. doi: 10.1007/s12149-024-02009-0. Epub 2024 Dec 14. PMID 39673015